CLINICAL TRIAL: NCT03411122
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Drug Interaction Potential of Napabucasin in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Drug Interaction Potential of Napabucasin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBI608-102
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Drug-drug Interactions
Keywords: Enzyme Inhibitors; Cytochrome P-450 Enzyme Inducers
MeSH Terms: interventions — napabucasin; Cytochrome P-450 Enzyme System

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single-sequence 3-period (Experimental): Period 1: napabucasin 240 mg BID on days 1-2 Period 2: cytochrome P450 probe drugs during days 1-4 Period 3: napabucasin 240 mg BID on days 1-11, cytochrome P450 probe drugs during days 6-9
  Interventions: Drug: napabucasin; Drug: cytochrome P450 (CYP450) probe drugs or BCRP transporter substrate

INTERVENTIONS:
Drug: napabucasin — Napabucasin will be administered at dose of 240 mg twice daily, every 12 hours (BID) on days 1-2 in period 1, and on days 1-11 in period 3.
  Other Names: BBI-608; BBI608
Drug: cytochrome P450 (CYP450) probe drugs or BCRP transporter substrate — CYP450 probe drugs or BCRP transporter substrate will be administered once every period during days 1-4 in period 2, and days 6-9 in period 3.

SUMMARY:
This is a phase I, single-center, open-label, single-sequence, 3-period, PK drug interaction study evaluating the effect of napabucasin in healthy volunteers on the single-dose PK of several cytochrome P450 (CYP450) probe drugs as well as a BCRP substrate.

ELIGIBILITY:
Inclusion Criteria

A subject will be eligible for inclusion in this study only if all the following criteria apply:

1. An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.
2. Subject is between the ages of 18 and 45 years, inclusive.
3. Subject is a female of childbearing potential with a negative pregnancy test or has documented surgical sterilization or is post-menopausal prior to Screening. All male and female subjects must agree to use contraception while participating in the study and for 30 days after their last dose of study drug unless surgically sterile or post-menopausal.. It is the Investigator's responsibility for determining whether the Subject has adequate birth control for study participation.
4. Subject has a body mass index between 18 and 34 kg/m^2 (weight/[height]^2).
5. Subject has normal (or abnormal and clinically insignificant according to the Investigator) laboratory values at screening.
6. Subject is medically normal with no significant abnormalities at the baseline physical examination.
7. Subject has the ability to understand the requirements of the study and a willingness to comply with all study procedures.
8. Subject has not consumed and agrees to abstain from taking any dietary supplements, herbal products, or non-prescription drugs (except as authorized by the Investigator and Medical Monitor) for 14 days prior to CRU admission through Follow-Up.
9. Subject has not consumed and agrees to abstain from taking any prescription drugs (except as authorized by the Investigator and Medical Monitor) during the 14 days prior to CRU admission through Follow-Up.
10. Subject has not consumed alcohol-containing beverages for 3 days prior to CRU admission and agrees not to consume alcohol through Follow-Up.
11. Subject has not consumed grapefruit, grapefruit juice, Seville oranges, and grapefruit- or Seville orange containing products within the 14 days prior to CRU admission and agrees not to consume grapefruit or grapefruit juice through Follow-Up.
12. Subject has not used tobacco- and nicotine-containing products within 2 months prior to the CRU admission and agrees to abstain from using tobacco- and nicotine-containing products through Follow-up.
13. Subject agrees to abstain from consuming caffeine- or chocolate-containing products from 3 days prior to CRU admission through Follow-up.

Exclusion Criteria

A Subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Subject has a history illicit drug abuse in the past year or current evidence of such abuse in the opinion of the Investigator.
2. Subject has positive findings on urine drug screen.
3. Subject is positive for human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C on Screening assessments.
4. Subject is determined to be a poor metabolizer for CYP2C19, CYP2C9 and/or CYP2D6.
5. Subject has a QTcF >450 msec (if male) or >470 msec (if female) at Screening.
6. Subject is pregnant or lactating.
7. Subject has an acute illness within 1 week of CRU admission.
8. Subject has a hypersensitivity or allergy to napabucasin or any of the probe drugs, or the ingredients of napabucasin or any of the probe drugs, or other clinically significant allergies.
9. Subject has donated plasma within 7 days of drug administration.
10. Subject has donated 1 or more pints of blood (or equivalent blood loss) within 30 days prior to drug administration.
11. Subject has a history of chronic Gastroesophageal reflux disease (GERD) or has used omeprazole or other proton pump inhibitors within 3 months of Screening.
12. Subject has participated in an investigational drug study within the 30 days prior to CRU admission.
13. Subject is an employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, or a family member of the employees or the Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics for napabucasin by assessing plasma concentration | Predose and up to 7 days post dose
Pharmacokinetics for probe drugs by assessing plasma concentration | Predose and up to 7 days post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Accel Research Sites, DeLand, Florida, United States

REFERENCES:
- [Derived] Dai X, Karol MD, Hitron M, Hard ML, Goulet MT, McLaughlin CF, Brantley SJ. Napabucasin Drug-Drug Interaction Potential, Safety, Tolerability, and Pharmacokinetics Following Oral Dosing in Healthy Adult Volunteers. Clin Pharmacol Drug Dev. 2021 Aug;10(8):824-839. doi: 10.1002/cpdd.961. Epub 2021 Jun 9. PMID 34107166